CLINICAL TRIAL: NCT04398212
Title: Visual and Ocular Sequelae of Computer Vision Syndrome: A Randomized Controlled Trial
Brief Title: Computer Vision Syndrome Visual Sequelae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Prof. Mohammed Iqbal, Assistant Professor of Ophthalmology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 5-10/4/2018
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Computer Vision Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-complaining group (Placebo Comparator): the students in this group are not complaining of CVS symptoms but will be examined to diagnose CVS or exclude it
  Interventions: Diagnostic Test: mfERG (multifocal-retinogram)
- Complaining group (Experimental): the students in this group are complaining of CVS symptoms but will be examined to document their complains and correlate to clinical findings
  Interventions: Diagnostic Test: mfERG (multifocal-retinogram)

INTERVENTIONS:
Diagnostic Test: mfERG (multifocal-retinogram) — mfERG will be performed for the students to document the effect of CVS on retina

SUMMARY:
the university students will respond to CVS-F3 survey form and then they will be subjected to complete ophthalmic examination and investigations

DETAILED DESCRIPTION:
CVS-F3 is a survey form consisted of up to 30 questions regarding Computer Vision Syndrome (CVS) complains, thereafter a randomized sample of students will be subjected to complete ophthalmic examination including visual acuity and refractive measurements, intraocular pressure measurements, Slitlamp and fungus examinations, mfERG examinations. the sudents will be requested to decrease their screen time and the examinations will be repeated one month later.

ELIGIBILITY:
Inclusion Criteria:

- University students

Exclusion Criteria:

* Amblyopia
* Anisometropia
* strabismus
* Previous eye surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 733 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
visual acuity | 1 month
  visual changes i.e. uncorrected distance visual acuity (UDVA) and corrected distance visual acuity (CDVA) using logMAR measurements following reduction of screen time
near vision | 1 month
  near vision changes following reduction of screen hours using card test, near visual acuity chart and near point test while the measurements will be diopters and lines of near chart

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Iqbal, MD. PhP, Principal Investigator — Sohag University
Locations (1):
- Faculty of medicine, Sohag, Egypt